CLINICAL TRIAL: NCT06965101
Title: Rapid Response MRI-Guided Palliative Radiotherapy
Brief Title: To Determine Whether it is Feasible to Treat Patients Requiring Urgent Radiotherapy Diagnosed With Metastatic Cord Compression (MSCC) on the Magnetic Resonance Linear Accelerator (MRL) in a Single Appointment and Compare it to the Standard of Care Radiotherapy Pathway
Acronym: RESONATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CFTSp246
Record Dates: First submitted 2025-04-11; First posted 2025-05-11 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Spinal Cord Compression
Keywords: Radiotherapy; MR Linac; MSCC; CT Sim Free; One Stop; MR Guided
MeSH Terms: conditions — Spinal Cord Compression

STUDY DESIGN:
Intervention Model Description: Non Randomised, single centre study design. Participants will choose, if they meet all eligibility criteria, which treatment group they would like to participate in. Either to receive Radiotherapy on the MR Linac or standard of care Radiotherapy.
  If participants do not meet the eligibility criteria and would like to participate they will be assigned to the standard of care Radiotherapy group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRL (Active Comparator): Using the MR Linac to deliver Radiotherapy in a single treatment without the need for a prior planning CT scan.
  Interventions: Radiation: Radiotherapy to the spine in a single appointment
- Standard of Care (Placebo Comparator): Using a conventional linear accelerator to deliver Radiotherapy in a single treatment, participants will require a prior planning CT appointment before Radiotherapy can be delivered.
  Interventions: Radiation: Radiotherapy to the spine in a single appointment

INTERVENTIONS:
Radiation: Radiotherapy to the spine in a single appointment — 8Gy/ 1# to be delivered to all participants using a single posterior direct field.

SUMMARY:
The goal of this clinical trial is to understand whether the Magnetic Resonance Linear Accelerator (MRL) could expedite Radiotherapy treatment for Metastatic Cord Compression (MSCC) by removing the need for a planning CT (pCT) scan prior to treatment. Radiotherapy will be delivered in one appointment on the MRL and compared to the standard of care of two appointments: a CT scan and a Radiotherapy appointment.

The main questions it aims to answer are:

* Can the MRL deliver successful treatment of MSCC in a single 1-hour appointment?
* Can the MRL treat participants within 24 hours from the doctor's decision to treat?
* Did it take less time from consent to completion of treatment when patients were treated on the MRL?
* Do the questionnaire scores reflect satisfaction with treatment on the MRL? Researchers will compare treatment on the MRL in one appointment to a group receiving standard of care radiotherapy in two appointments.

Participants in both groups will receive the same prescription of 8Gray (Gy) in one treatment (fraction) delivered with one posterior-anterior beam as per our department policies and national standards.

Participants will be asked to complete an optional questionnaire prior to treatment to monitor the diversity of the study population. This questionnaire is anonymised, no personal data that could identify a participant is collected on this questionnaire.

After treatment participants will be asked to complete an experience questionnaire, to assess treatment experience.

Once the questionnaire is complete active participation in the trial is no longer needed, researchers will monitor participants notes for up to 12 months after treatment to record participant well being and function.

DETAILED DESCRIPTION:
Metastatic cord compression occurs in 5-10% of patients with cancer often affected the ends stages of a patient's illness. The benefit of palliation is directly related to the speed of treatment, National Institute of Health and Care Excellence (NICE) guidelines recommend that radiotherapy is given within 24 hours of a decision to treat. A recent audit of the current referrals and pathway showed the average time from consultation to treatment is 2.10 days (SD 12.2 days). This audit concluded the need to improve the speed of access to care.

The current pathway includes a scan for diagnosis (MRI), a visit for a planning CT and time to plan the treatment before treatment delivery. This can take many hours or even days. To provide quicker access to care it is intended to use the MR Linac with an integrated adaptive radiotherapy platform, to deliver a scan, plan and treat model in a single appointment.

Preliminary work has modelled dose differences due to the presence of a magnetic field, known as the electron return effect and developed an MR only workflow using a simple planning technique to enable the online scan, plan and treat model.

The primary objective is to test the feasibility of a one-stop MR guided palliative radiotherapy programme for patients with MSCC.

Secondary objectives are:

* To reduce overall time from decision to treat to treatment delivery.
* Reduce the number of appointments and procedure required to provide palliative radiotherapy for patients with MSCC.
* Compare participant experience of MSCC treatment on the MR Linac to the current standard of care pathway.

This is a single centre, non-randomised clinical trial. All patients referred for radiotherapy to treat MSCC who can provide informed consent can be considered. Participants will be asked to have treatment on the MR Linac within a single appointment and complete an experience questionnaire. If participants would not like to have treatment on the MRL or do not meet the inclusion criteria participants can continue the standard of care pathway with the addition of completing an experience questionnaire and the data and answers will be used for analysis. If patients would not like to participate, standard of care radiotherapy will be delivered and this patient data will not be used for this study.

The study is expected to recruit up to 72 participants over a 2-year period using a 1:2 ratio. Up to 24 participants will be recruited to the MR Linac Arm of the study. This sample is based on resource constraints, the MR Linac can accommodate one patient per month on average. Recruitment will be a 1:2 ratio to reduce bias to the investigational arm.

To test the aim, to improve the speed of access of care, timings will be collected at certain time points throughout the pathway:

* Clinical decision to treat the participant
* Time of treatment consent
* Time of Radiotherapy Planning scan (Standard of Care only)
* Time of Radiotherapy Completion

The study will consist of:

1. MSCC team confirm diagnosis & organise for the patient to be transferred to the Christie. (Day 0)
2. Referral to Radiotherapy (Day 0)
3. Approached in person by the Research Team & MRI screening. (Day 1)
4. Consent to Radiotherapy. (Day 1)
5. Consent to Study. (Day 1)
6. Optional Equality diversity and inclusivity (EDI) Questionnaire completed. (Day1)
7. Patient prepared in MRL clinical system or given RTP appointment. (Day 1)
8. Radiotherapy treatment on MRL or Conventional Linac. (Day 1 -7)
9. Patient experience questionnaire completed. (Same day as treatment)
10. Patient outcomes will be determined from clinical notes. (1,3,6,12 months following treatment)

A participant is free to withdraw from the clinical trial at any point without giving a reason.

This study will run for 3 years in total, 2 years for recruitment plus one year for follow up unless early termination is required.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Diagnosis of MSCC
* Referred for an 8Gy, Single Fraction of Radiotherapy
* 18 years or older.
* Able to give informed consent in writing or verbally.
* Willing to complete patient experience questionnaire
* Willing to have the research team review their case notes for up to 1 year following

Exclusion Criteria:

* Participant does not have capacity and cannot give informed consent.
* Any evidence of significant clinical disorder or laboratory finding which, in the opinion of the investigator, make it undesirable for the patient to participate in the study.
* Participant is unwilling to allow researchers to access their clinical notes and diagnostic scans.
* Participant is unwilling to complete an experience questionnaire
* The participant cannot speak or understand English.

Exclusion Criteria MRL arm:

* Any contraindications to MRI identified after MRI safety screening
* Unable to tolerate MRI scanning
* Uncontrolled pain/ poor pain control.
* MSCC in the cervical spine.
* More than one vertebral level of compression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-11-04 (Estimated); Study Completion 2028-11-04 (Estimated)

PRIMARY OUTCOMES:
Successful treatment of Metastatic Spinal Cord Compression in a single 1 hour appointment for 80% of patients on the MRL Arm | The event is assessed on a single day (within 24hours) over a single appointment. From the time the patient enters the treatment room to the time the radiotherapy beam is completed (Up to 2 hours in length).
  "Successful treatment" is defined as the complete delivery of the Radiotherapy treatment beam to the area of Metastatic Spinal Cord Compression.
  The measurement used to assess appointment length will be time, recorded in hours, minutes and seconds. Time from the patient entering the room to the treatment beam completing.

SECONDARY OUTCOMES:
80% of patients on the MRL Arm treated within 24 hours from decision to treat | From clinician's referral to the completion of the treatment beam (Assessed for up to 7 days).
  The measurement used to assess will be the length of time (in days, hours, minutes). Assessed from the time the Radiotherapy referral form is submitted by the clinician to when the Radiotherapy treatment beam is completed.
80% of patients on the MRL Arm spend less time from consent to completion of treatment when compared to the Standard of Care Arm | From time of treatment consent to completion of the treatment beam (Assessed for up to 7 days)
  The measurement used to assess will be the length of time (in days, hours, minutes). Assessed from the time the Radiotherapy treatment consent form is signed by the participant to when the Radiotherapy treatment beam is completed.
80% of the MRL Arm questionnaire scores reflect satisfaction with the treatment | After completion of Radiotherapy (Within 2 hours of the treatment beam being completed)
  The experience questionnaire collects answers on a 4-point Likert scale from 0-3. "Satisfaction" is defined as scores that are above 1 for positive questions, those that high scores indicate a positive experience. Or scores that are below 2 for negative questions, those that high scores indicate a negative experience.
The study population is representative of the population referred for Radiotherapy for Metastatic Spinal Cord Compression. | At the time of enrolment (within 2 hours of signing consent form)
  Voluntary questionnaire completed. Equality Diversity and Inclusion (EDI) data from this study will be compared to local and national EDI data statistics for MSCC patients. The percentage of characteristics represented in the study compared to the wider population.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia L Eccles, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data for this study will be pseudo-anonymised and kept securely at The Christie, only accessible to those employed by the Christie NHS Foundation Trust.
  Due to the data not being fully anonymised and to preserve patient confidentiality the data from this study will not be shared.

REFERENCES:
- [Background] Olausson K, Holst Hansson A, Zackrisson B, Edvardsson D, Ostlund U, Nyholm T. Development and psychometric testing of an instrument to measure the patient's experience of external radiotherapy: The Radiotherapy Experience Questionnaire (RTEQ). Tech Innov Patient Support Radiat Oncol. 2017 Jul 24;3-4:7-12. doi: 10.1016/j.tipsro.2017.06.003. eCollection 2017 Sep-Dec. PMID 32095560
- [Background] Barnes H, Alexander S, Bower L, Ehlers J, Gani C, Herbert T, Lawes R, Moller PK, Morgan T, Nowee ME, Smith G, van Triest B, Tyagi N, Whiteside L, McNair H. Development and results of a patient-reported treatment experience questionnaire on a 1.5 T MR-Linac. Clin Transl Radiat Oncol. 2021 Jun 29;30:31-37. doi: 10.1016/j.ctro.2021.06.003. eCollection 2021 Sep. PMID 34307911
- [Background] Hales RB, Rodgers J, Whiteside L, McDaid L, Berresford J, Budgell G, Choudhury A, Eccles CL. Therapeutic Radiographers at the Helm: Moving Towards Radiographer-Led MR-Guided Radiotherapy. J Med Imaging Radiat Sci. 2020 Sep;51(3):364-372. doi: 10.1016/j.jmir.2020.05.001. Epub 2020 Jun 26. PMID 32600981
- [Background] Benson R, Clough A, Nelder C, Pitt E, Portner R, Vassiliou M, McDaid L, Choudhury A, Rembielak A, Eccles C. Evaluation of the palliative radiotherapy pathway in a single institute: Can an MR Linac improve efficiency? J Med Imaging Radiat Sci. 2022 Jun;53(2 Suppl):S44-S50. doi: 10.1016/j.jmir.2021.11.010. Epub 2021 Dec 16. PMID 34922879
- See also: NICE Guideline NG234 - Spinal Metastasis and Metastatic Spinal Cord Compression — https://www.nice.org.uk/guidance/ng234/chapter/Recommendations#radiotherapy